CLINICAL TRIAL: NCT06346262
Title: Seizure Rescue Medication (RM) as Part of a Comprehensive Epilepsy Self-management Package of Care
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Principal Investigator, Martha Sajatovic, Physician, UHMG, University Hospitals Cleveland Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STUDY20230921
Record Dates: First submitted 2024-03-22; First posted 2024-04-04 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Epilepsy
Keywords: Epilepsy Self Management; Epilepsy; Seizure; Reduction medication; Anti-seizure medication
MeSH Terms: conditions — Epilepsy; Seizures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- SMART RM (Experimental): The SMART-RM will consist of 8 group-format, 45-60 minute sessions (up to 11 participants per group), which will be collaboratively delivered by a Nurse Educator (NE) and a Peer Educator (PE). The intervention will be remotely delivered in a web-based format using a secure web teleconferencing system (such as Zoom) that will allow us to set up a virtual meeting room. Following the group-session series, participants will have 3 monthly telephone maintenance sessions lasting around 15 minutes. Maintenance session web/telephone calls will be made to study participants by a NE with experience in epilepsy and/or chronic health condition management.
  Interventions: Behavioral: SMART RM; Drug: Valtoco Nasal Product

INTERVENTIONS:
Behavioral: SMART RM — The SMART-RM will consist of 8 group-format, 45-60 minute sessions (up to 11 participants per group), which will be collaboratively delivered by a Nurse Educator (NE) and a Peer Educator (PE).
Drug: Valtoco Nasal Product — Medication dosing will follow recommendations in the Valtoco package insert and managed by the epilepsy clinician.

SUMMARY:
This study will be done in two phases. Using stakeholder input (community advisory board (CAB)), the study team will adapt the SMART program to incorporate education and self-management support for use of Rescue Medication (RM) to manage seizure occurrence among Persons With Epilepsy (PWE) who have repetitive seizures. Additional content/support materials, pending input stakeholder might include posters/hand-outs that present information on the use of RM in a way that is engaging and salient to PWE. It is expected that participants will be in Phase 1 for about 3 months and participate in the CAB 2 or 3 times via zoom for 60-90 minutes/meeting. The advisory board will provide input on needed refinement of an adapted version of SMART based on their individual experiences. It is anticipate the total time commitment to be no more than 6 hours over 3 months, spread out over 2-3 meetings with review of materials possible in between meetings.

Phase 2: The investigators will use a 6-month prospective trial design to test engagement with and effects of SMART-RM among approximately 35 adult (≥ 18 years) PWE who have repetitive seizures.

ELIGIBILITY:
Inclusion Criteria:

Phase 1 Patient with epilepsy inclusion criteria:

* Have epilepsy
* Have experience with RM
* Be 18 years or older
* Be able to speak and understand English
* Be able to provide written, informed consent to study participation

Phase 1 Caregiver inclusion criteria

* Provide care support to an individual with epilepsy
* Be 18 years or older
* Be able to speak and understand English
* Be able to provide written, informed consent to study participation

Phase 1 Provider inclusion criteria

* Provide care for individuals with epilepsy - this may include (not limited to) physician, nurse practitioner, physician assistant, nurse, social worker, psychologist
* Be 18 years or older
* Be able to speak and understand English
* Be able to provide written, informed consent to study participation

Inclusion criteria for PEs:

* Have epilepsy
* Have experience with RM
* Be 18 years or older
* Be able to speak and understand English
* Be able to provide written, informed consent to study participation

Inclusion criteria for participants who will receive SMART-RM:

* Have received a previous diagnosis of epilepsy
* Be adults ≥ age 18,
* While on a regimen of anti-epileptic medication, still be experiencing bouts of seizures (e.g. frequent break through or acute repetitive seizures) distinct from their usual seizure pattern , and, in the opinion of the study epilepsy clinician, may need benzodiazepine intervention for seizure control
* Have experienced at least 3 seizures but not more than 100 seizures in the previous 6 months. If there have only been 3 seizures in the last 6 months, two of the seizures should be within approximately 24 hours of each other (not more than 48 hours apart)
* Be able to speak and understand English
* Be able to provide written, informed consent to study participation

Exclusion Criteria:

Exclusion criteria for participants who will receive SMART-RM:

* Individuals who have had allergic reaction to diazepam or who have medical/psychiatric that are contraindications to the use of diazepam
* Individuals prescribed opioid medications
* Individuals with acute narrow angle glaucoma
* Individuals with known dependence on benzodiazepines or current benzodiazepine abuse.
* Actively suicidal/homicidal
* Individuals with a diagnosis of dementia
* Individuals who are unable to provide written informed consent to participate in study and who do not have a legally authorized representative or individuals who are unable to participate in study procedures.
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-03-05 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in number of seizures as measured by patient report. | Baseline, 6 months

SECONDARY OUTCOMES:
Change in quality of life as measure by QOLIE-31 | Baseline, 10 week, 24 week
  Quality of life (QOL) will be assessed using the QOLIE-31, a validated tool to assess quality of life specifically in people with epilepsy with higher numbers reflecting a more favorable health state.
Change in functional status as measure by Short-Form Health Survey (SF-36) | Baseline, 10 week, 24 week
  Functional status will be assessed using the 36-item Short-Form Health Survey (SF-36), a multipurpose, short-form health survey with 36 questions that yields two psychometrically based components: a physical component summary and mental component summary. Scores range from 0 (worst functioning) to 100 (best functioning). The SF-36 is a generic measure of functional health status and has proven useful for comparing the relative burden of diseases.
Change in depressive symptoms as measure by Patient Health Questionnaire (PHQ-9) | Baseline, 10 week, 24 week
  Depressive symptom severity will be assessed using the nine- item Patient Health Questionnaire (PHQ-9), a widely used and validated self-rated depression scale. The PHQ-9 incorporates Diagnostic and Statistical Manual of Mental Disorders diagnostic criteria, with scores ranging from 0 to 27. Higher scores indicate worse depression severity. The PHQ-9 has been widely used to measure depressive symptom severity in epilepsy.
Change in epilepsy self management as measure by Epilepsy Self-Efficacy Scale (ESES) | Baseline, 10 week, 24 week
  Self-efficacy will be measured using the 33-item Epilepsy Self-Efficacy Scale (ESES), with scores ranging from 0 to 330 and higher scores indicating better self-efficacy. Social support will be measured with the 12-item.
Change in epilepsy self management as measure by Multidimensional Scale of Perceived Social Support (MSPSS) | Baseline, 10 week, 24 week
  Multidimensional Scale of Perceived Social Support (MSPSS), which measures perception of social support provided by family and friends, as well as satisfaction with that support. The MSPSS score ranges from 1 to 84, with higher scores indicating better social support.
Change in epilepsy self management as measure by Epilepsy Self-Management Scale (ESMS) | Baseline, 10 week, 24 week
  Overall epilepsy self-management competency will be measured using the Epilepsy Self-Management Scale (ESMS); scores range from 1 to 190, with higher scores indicating better self-management of epilepsy.
Change in epilepsy self management as measure by Epilepsy Stigma Scale (ESS) | Baseline, 10 week, 24 week
  Stigma for epilepsy will be measured using the Epilepsy Stigma Scale (ESS) In the ESS, scores range from 7 to 70; each item is rated on a 7-point scale from strongly disagree to strongly agree, with higher numbers indicating greater perceived stigma
Change in number of emergency room visit as measure by patient report | Baseline, 10 week, 24 week
Change in number of hospitalizations as measure by patient report | Baseline, 10 week, 24 week
Change in number of non study outpatient services utilization as measure by patient report | Baseline, 10 week, 24 week

CONTACTS AND LOCATIONS:
Overall Officials: Martha Sajatovic, MD, Principal Investigator — University Hospitals
Locations (1):
- University Hospitals Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No